CLINICAL TRIAL: NCT00366405
Title: Comparison of the Torsional Handpiece to Conventional Handpiece During Routine Phacoemulsification
Status: Completed | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Kerry D. Solomon, Medcial University of South Carolina
Other Study IDs: MRC-06-001
Record Dates: First submitted 2006-08-17; First posted 2006-08-21 (Estimated); Last update posted 2010-10-04 (Estimated); Status verified 2010-10

CONDITIONS: Cataract Extraction
Keywords: cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate the visual outcomes, amount of inflammation, endothelial cell loss, and the efficiency of a torsional handpiece compared to a conventional handpiece during surgery to remove your cataracts.

DETAILED DESCRIPTION:
With the introduction of new phaco-emulsification systems, the cataract surgery has become a very safe procedure. The new machines combine fewer surges, lower amount of ultrasound and more controlled anterior chamber depth, as well as lower incidence of thermal burns of the incision site.1-4

Alcon's Infiniti Vision System phacoemulsification machine includes now a torsional handpiece (OZiL™). The goal of OZiL™ is to minimize the surgery impact by reducing temperature increase, turbulence and incision stress. This handpiece has a sideways movement that does not repel the cataract during its extraction making the removal more continuous, maintains occlusion which facilitates vacuum build-up and reduces flow through the anterior chamber decreasing turbulence, therefore reducing the likelihood of lens particles damaging the corneal endothelial cells.

The purpose of this study is to compare visual outcomes, induction of inflammation, endothelial cell loss and efficiency of the torsional handpiece vs. the conventional phacoemulsification handpiece when using the Alcon Infiniti Vision System.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral senile cataracts.
* Cataract density up to 3+.
* 50 years of age or older.
* Patient must desire cataract extraction.
* Expected maximum of 4 weeks and minimum of 1 week interval between first and second eye surgeries.
* Willing and able to comply with scheduled visits and other study procedures.

Exclusion Criteria:

* Preoperative ocular pathology: amblyopia, rubella cataract, proliferative diabetic retinopathy, macular edema, retinal detachment, uveitis, history of iritis, iris neovascularization, medically uncontrolled glaucoma, microphthalmus or macrophthalmus, optic nerve atrophy, macular degeneration with visual acuity of less than 20/40, glaucoma with the presence of visual field defects
* Corneal irregularities potentially affecting visual acuity: keratoconus, corneal dystrophy, corneal opacities.
* Low endothelial cell count (less than 1500 cells/mm2)
* Any concurrent infectious/non infectious conjunctivitis, keratitis or uveitis in either eye.
* Any clinically significant, serious or severe medical or psychiatric condition.
* Participation in (or current participation) any investigational drug or device trial within the previous 30 days prior to the start date of this trial.
* Previous intraocular or corneal surgery.
* Other ocular surgery at the time of the cataract extraction.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Bilateral senile cataracts. Cataract density up to 3+. 50 years of age or older. Patient must desire cataract extraction. Expected maximum of 4 weeks and minimum of 1 week interval between first and second eye surgeries.
  Willing and able to comply with scheduled visits and other study procedures.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2006-02; Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kerry D Solomon, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Storm Eye Institute, Medical University of South Carolina, Charleston, South Carolina, United States